CLINICAL TRIAL: NCT02288468
Title: One Pass thalamIc aNd subthalamIc stimulatiON
Acronym: OPINION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Volker Arnd Coenen, Prof. Dr., University Hospital Freiburg
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P000568; DRKS00007526 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2014-11-03; First posted 2014-11-11 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STN (Experimental): Deep Brain Stimulation of Nucleus subthalamicus with Vercise™ Deep Brain Stimulation System.
  The STN will be typically reached with the most distal contacts of the DBS electrode (8 contact). Imaging studies (postop helical CT and re-fusion to planning MRI data) will allow for the identification of contacts located in the STN. We expect the STN to be typically covered by contacts 1-4 of the Vercise™ DBS lead. Typically, only the most superficial contacts (3,4) will be activated after a monopolar review of each contact. In this monopolar review the therapeutic widths of each contact will be tested for its effectiveness in tremor reduction, reduction of rigidity and bradykinesia. Typical settings will be: Frequency 130-180 Hz, pulse width 60-90 us, Amplitude 1-7 mA.
  Interventions: Device: Vercise™ Deep Brain Stimulation System
- Vim/DRT (Experimental): Deep Brain Stimulation of Ventral intermediate nucleus with Vercise™ Deep Brain Stimulation System.
  The thalamic target (Vim/DRT) will be typically reached with the proximal contacts. Imaging studies (postop helical CT and re-fusion to planning MRI data) will allow for the identification of contacts located the thalamic target. We expect the thalamic target to be typically covered by contacts 5-8 of the Vercise™ DBS lead. We will perform a monopolar review of each contact. In this monopolar review the therapeutic widths of each contact will be tested for its effectiveness in tremor reduction and the occurrence of side effects (typically capsular e.g. facial contraction). Typical settings will be: Frequency 130-180 Hz, pulse width 60-90 us, Amplitude 1-7 mA.
  Interventions: Device: Vercise™ Deep Brain Stimulation System
- STN+Vim/DRT (Experimental): Combined Deep Brain Stimulation of Nucleus subthalamicus and Ventral intermediate nucleus with Vercise™ Deep Brain Stimulation System.
  STN+Vim/DRT stimulation is essentially a combination of the previously described procedure.
  Interventions: Device: Vercise™ Deep Brain Stimulation System

INTERVENTIONS:
Device: Vercise™ Deep Brain Stimulation System — The Vercise™ DBS System includes a Stimulator with DBS Leads for unilateral or bilateral stimulation. There are also DBS Extensions that allow the DBS Leads mounted in the skull to be extended to reach the Stimulator implanted near the clavicle.
  The rechargeable Vercise DBS System utilizes current steering across eight contacts per DBS Lead to provide precise positioning of stimulation. The Stimulator is controlled by a handheld Remote Control, and can be interfaced with a Clinician's Programmer using the Bionic Navigator™ Software. Periodically, the Stimulator battery must be replenished with an RF (radiofrequency) charging device provided in the Patient DBS Charging Kit.
  Other Names: Vercise DBS

SUMMARY:
Main part of the study:

Randomised, active controlled, double blinded (patient and observer blinded), monocentric trial with three treatments, three periods and six treatment sequences allocated according to a Williams design

Open Label Extension:

After study treatment as described above, patients will be treated unblinded in their preferred stimulation mode until 36 months after implantation.

DETAILED DESCRIPTION:
Tremor is the most salient symptom of Parkinson's disease (IPS=idiopathic Parkinson syndrome). Other symptoms are bradykinesia, rigidity and postural instability. As much as 75% of patients with IPS show resting tremor. Initially, tremor is typically unilateral and only visible in stress situation. In the later stage of the disease it becomes bilateral. The OPINION trial aims at the investigation of a combined approach to thalamic/subthalamic deep brain stimulation (DBS) for the treatment of patients with tremor dominant IPS or patients with equivalent type IPS who perceive tremor to be their dominant symptom. The planned approach will for the first time allow for the direct comparison of each condition in a homogeneous patient population and will furthermore allow an intra-individual comparison of the different stimulation conditions (Ventral intermediate nucleus (Vim/DRT) - Subthalamic nucleus (STN) - Vim/DRT+STN) with the outcome parameter "quality of life".

Patients will be registered to the trial and will undergo screening procedures (for eligibility criteria please see Inclusion and Exclusion criteria). If the patient is eligible the Investigational Medical Device (IMD) will be implanted (which is the Vercise™ Deep Brain Stimulation System manufactured by Boston Scientific). After implantation the IMD will remain OFF for a period of 1 month.

1 month after implantation treatment will be started. Patients will be randomized to one of the following 3 treatment groups: Subthalamic nucleus (STN) or Ventral intermediate nucleus (Vim/DRT) or combined stimulation (Vim/DRT+STN). Patients will undergo all three treatment groups each lasting 3 months. The patient is blinded meaning that study patients will not know what kind of treatment (e.g. mode/region of stimulation) they receive.

10 months after implantation the final visit of the randomized study will be performed. After that, patients will be asked to take part in an open label extension phase of the study where they will be treated unblinded according to established guidelines and according to their own preferred stimulation mode, just as they would be in a clinical routine setting. The extension phase is concluded by an end of study visit at 36 months after implantation.

After the end of the trial, further treatment will be performed at the Department of Stereotactic and Functional Neurosurgery in Freiburg (Germany) according to established guidelines. Devices will be monitored 3-6 monthly Patient's medications will be adjusted as to the level of best treatment adjunct to stimulation.

Study endpoints (e.g. quality of life) will be evaluated by a blinded rater. In addition, an external video rating will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 35 and ≤ 75 years with a life expectancy of at least 5 years
2. Patients with Parkinson's disease according to the criteria of the British Brain Bank as diagnosed by an in movement disorder specialized neurologist
3. Parkinson patients are included with a medical treatment resistant and disabling resting and/or postural tremor as their major complaint and with a less prominent or absent hypokinetic-rigid component of their disease.
4. Absence of postural instability (which would be aggravated under STN DBS)
5. Hoehn & Yahr stage 1-3. After stadium 3 patients will show increased incidence of falling that can be aggravated by (typical) STN DBS
6. Disease duration for at least 2 years and routine DAT-scan shows clear indication for Parkinsonism and atypical Parkinson syndromes are ruled out by routine glucose (FDG) PET
7. PDQ-39 to be completed within 42 days prior surgery
8. Written informed consent

Exclusion Criteria:

1. Major Depression with suicidal thoughts
2. Dementia (Mattis Dementia Rating Score ≤ 130)
3. Patients with lifetime primary psychotic disorder, schizophrenia, or schizoaffective disorder
4. Patients with acute psychosis as diagnosed by a psychiatrist
5. Nursing care at home
6. Unable to give written informed consent
7. Surgical contraindications like deformed or displaced or not discernable target region, scarring after brain disease (infarction), need for continuous anticoagulation that cannot be bridged in order to obtain normal coagulation
8. Patients with advanced stage cardiovascular disease
9. Patients under immunosuppressive or chemotherapy because of malignant disease
10. Patients who had previous intracranial surgery
11. Patients who are already under DBS therapy
12. Patients with aneurysm clips
13. Patients with cochlear implants
14. Simultaneous participation or previous participation within 30 days prior to start of screening in a clinical trial involving investigational medicinal product(s) or investigational medical device(s)
15. Medications that are likely to cause interactions in the opinion of the investigator
16. Known or persistent abuse of medication, drugs or alcohol
17. Persons who are in a relationship of dependence/employment with the sponsor or the investigator
18. Fertile women not using adequate contraceptive methods: female condoms, diaphragm or coil, each used in combination with spermicides; intra-uterine device; hormonal contraception in combination with a mechanical method of contraception;
19. Current or planned pregnancy, nursing period
20. Contraindications according to device instructions or Investigator's Brochure:

    * Diathermy: Shortwave, microwave, and/or therapeutic ultrasound diathermy. The energy generated by diathermy can be transferred to the Vercise™ DBS System, causing tissue damage at the contact site resulting in severe patient injury or death.
    * Magnetic Resonance Imaging (MRI): Patients implanted with the Vercise™ DBS System should not be subjected to MRI.
    * Patient incapability: Patients who are unable to properly operate the Remote Control and Charging System should not be implanted with the Vercise™ DBS System.
    * Poor surgical risks: The Vercise™ DBS System is not recommended for patients who - because of their primary disease or additional co-morbidities - are not likely to benefit from the DBS system implantation.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Change in PDQ-39 total score | From baseline every 3 months up to 9 months
  Change in PDQ-39 total score from base value (i.e. mean value of screening and baseline visit) until end of each treatment (Vim/DRT-DBS, STN-DBS, combined STN+Vim/DRT-DBS) 3 months after start of each treatment up to 9 months

SECONDARY OUTCOMES:
Change in FTMTRS | From baseline every 3 months up to 9 months, and at 36 months
  Change in Fahn-Tolosa-Marin Tremor Rating Scale (FTMTRS) every three months after start of each treatment (Vim/DRT-DBS, STN-DBS, combined STN+Vim/DRT-DBS), and at 36 months, compared to base value (i.e. mean value of screening and baseline visit)recording at the tremor peak in tremor analysis
Change in UPDRS motor score (part III, except items 20 & 21) | From baseline every 3 months up to 9 months, and at 36 months
  Change in Unified Parkinson's Disease Rating Scale (UPDRS) motor score (part III, except items 20 & 21) every three months after start of each treatment (Vim/DRT-DBS, STN-DBS, combined STN+Vim/DRT-DBS), and at 36 months, compared to base value (i.e. mean value of screening and baseline visit)
Change in UPDRS (part III, tremor subscore (items 20 & 21)) or total power of accelerometry recording at the tremor peak in tremor analysis | From baseline every 3 months up to 9 months, and at 36 months
  Change in UPDRS (part III, tremor subscore (items 20 & 21)) or total power of accelerometry recording at the tremor peak in tremor analysis every three months after start of each treatment (Vim/DRT-DBS, STN-DBS, combined STN+Vim/DRT-DBS), and at 36 months, compared to base value (i.e. mean value of screening and baseline visit)
Clinical Global Impression Scale (CGI-I) | Screening, baseline, then every 3 months until month 10, and at 36 months
  Assessment of Clinical Global Impression Scale (CGI-I) at screening, at baseline (month 1) and then every three months after start of each treatment (Vim/DRT-DBS, STN-DBS, combined STN+Vim/DRT-DBS) until month 10, and at 36 months
Change in PDQ-39 total score at 36 months | Baseline, month 36
  Change in PDQ-39 total score from base value (i.e. mean value of screening and baseline visit) until 36 months after implantation
Psychiatric assessment: C-SSRS | Screening, baseline, then every 3 months until month 10, and at 36 months
  Psychiatric assessment: Columbia Suicide Severity Rating Scale (C-SSRS) at screening, at baseline (month 1) and then every three months after start of each treatment (Vim/DRT-DBS, STN-DBS, combined STN+Vim/DRT-DBS) until month 10, and at 36 months
Psychiatric assessment: YMRS | Screening, baseline, then every 3 months until month 10, and at 36 months
  Psychiatric assessment: Young Mania Rating Scale (YMRS) at screening, at baseline (month 1) and then every three months after start of each treatment (Vim/DRT-DBS, STN-DBS, combined STN+Vim/DRT-DBS) until month 10, and at 36 months
Psychiatric assessment: MADRS | Screening, baseline, then every 3 months until month 10, and at 36 months
  Psychiatric assessment: Montgomery-Asberg Depression Scale (MADRS) at screening, at baseline (month 1) and then every three months after start of each treatment (Vim/DRT-DBS, STN-DBS, combined STN+Vim/DRT-DBS) until month 10, and at 36 months
Psychiatric assessment: BIS-11 | Screening, baseline, then every 3 months until month 10, and at 36 months
  Psychiatric assessment: Barratt Impulsiveness Scale (BIS-11) at screening, at baseline (month 1) and then every three months after start of each treatment (Vim/DRT-DBS, STN-DBS, combined STN+Vim/DRT-DBS) until month 10, and at 36 months
Assessment of (Serious) Adverse Events related to Investigational Medical Device, surgical procedures, stimulation settings and/or changes to medication | Starting from implantation of device until last visit at month 36
  Assessment of Adverse Events (AEs) and Serious Adverse Events (SAEs) related to Investigational Medical Device (IMD), surgical procedures, stimulation settings and/or surgical procedures

CONTACTS AND LOCATIONS:
Overall Officials: Volker Coenen, MD, Principal Investigator — University Hospital Freiburg
Locations (1):
- University of Freiburg - Medical Center - Dept. of Stereotactic and Functional Neurosurgery, Freiburg im Breisgau, Germany

REFERENCES:
- [Background] Hilker R, Benecke R, Deuschl G, Fogel W, Kupsch A, Schrader C, Sixel-Doring F, Timmermann L, Volkmann J, Lange M; German Deep Brain Stimulation Association. [Deep brain stimulation for Parkinson's disease. Consensus recommendations of the German Deep Brain Stimulation Association]. Nervenarzt. 2009 Jun;80(6):646-55. doi: 10.1007/s00115-009-2695-3. German. PMID 19360386
- [Background] Limousin P, Speelman JD, Gielen F, Janssens M. Multicentre European study of thalamic stimulation in parkinsonian and essential tremor. J Neurol Neurosurg Psychiatry. 1999 Mar;66(3):289-96. doi: 10.1136/jnnp.66.3.289. PMID 10084526
- [Background] Rehncrona S, Johnels B, Widner H, Tornqvist AL, Hariz M, Sydow O. Long-term efficacy of thalamic deep brain stimulation for tremor: double-blind assessments. Mov Disord. 2003 Feb;18(2):163-70. doi: 10.1002/mds.10309. PMID 12539209
- [Background] Krack P, Pollak P, Limousin P, Benazzouz A, Benabid AL. Stimulation of subthalamic nucleus alleviates tremor in Parkinson's disease. Lancet. 1997 Dec 6;350(9092):1675. doi: 10.1016/s0140-6736(97)24049-3. No abstract available. PMID 9400514
- [Background] Volkmann J, Daniels C, Witt K. Neuropsychiatric effects of subthalamic neurostimulation in Parkinson disease. Nat Rev Neurol. 2010 Sep;6(9):487-98. doi: 10.1038/nrneurol.2010.111. Epub 2010 Aug 3. PMID 20680036
- [Background] Fraix V, Pollak P, Moro E, Chabardes S, Xie J, Ardouin C, Benabid AL. Subthalamic nucleus stimulation in tremor dominant parkinsonian patients with previous thalamic surgery. J Neurol Neurosurg Psychiatry. 2005 Feb;76(2):246-8. doi: 10.1136/jnnp.2003.022707. PMID 15654041
- [Background] Deuschl G, Schade-Brittinger C, Krack P, Volkmann J, Schafer H, Botzel K, Daniels C, Deutschlander A, Dillmann U, Eisner W, Gruber D, Hamel W, Herzog J, Hilker R, Klebe S, Kloss M, Koy J, Krause M, Kupsch A, Lorenz D, Lorenzl S, Mehdorn HM, Moringlane JR, Oertel W, Pinsker MO, Reichmann H, Reuss A, Schneider GH, Schnitzler A, Steude U, Sturm V, Timmermann L, Tronnier V, Trottenberg T, Wojtecki L, Wolf E, Poewe W, Voges J; German Parkinson Study Group, Neurostimulation Section. A randomized trial of deep-brain stimulation for Parkinson's disease. N Engl J Med. 2006 Aug 31;355(9):896-908. doi: 10.1056/NEJMoa060281. PMID 16943402
- [Background] Okun MS, Rodriguez RL, Foote KD, Sudhyadhom A, Bova F, Jacobson C, Bello B, Zeilman P, Fernandez HH. A case-based review of troubleshooting deep brain stimulator issues in movement and neuropsychiatric disorders. Parkinsonism Relat Disord. 2008 Nov;14(7):532-8. doi: 10.1016/j.parkreldis.2008.01.001. Epub 2008 Mar 5. PMID 18325819
- [Background] Coenen VA, Allert N, Paus S, Kronenburger M, Urbach H, Madler B. Modulation of the cerebello-thalamo-cortical network in thalamic deep brain stimulation for tremor: a diffusion tensor imaging study. Neurosurgery. 2014 Dec;75(6):657-69; discussion 669-70. doi: 10.1227/NEU.0000000000000540. PMID 25161000
- [Background] LANCE JW, SCHWAB RS, PETERSON EA. Action tremor and the cogwheel phenomenon in Parkinson's disease. Brain. 1963 Mar;86:95-110. doi: 10.1093/brain/86.1.95. No abstract available. PMID 13928399
- [Background] Coenen VA, Prescher A, Schmidt T, Picozzi P, Gielen FL. What is dorso-lateral in the subthalamic Nucleus (STN)?--a topographic and anatomical consideration on the ambiguous description of today's primary target for deep brain stimulation (DBS) surgery. Acta Neurochir (Wien). 2008 Nov;150(11):1163-5; discussion 1165. doi: 10.1007/s00701-008-0136-x. Epub 2008 Oct 29. PMID 18958389
- [Background] Zrinzo L, Holl EM, Petersen EA, Limousin P, Foltynie T, Hariz MI. Skewering the subthalamic nucleus via a parietal approach. Stereotact Funct Neurosurg. 2011;89(2):70-5. doi: 10.1159/000323371. Epub 2011 Feb 2. PMID 21293165
- [Background] Coenen VA, Allert N, Madler B. A role of diffusion tensor imaging fiber tracking in deep brain stimulation surgery: DBS of the dentato-rubro-thalamic tract (drt) for the treatment of therapy-refractory tremor. Acta Neurochir (Wien). 2011 Aug;153(8):1579-85; discussion 1585. doi: 10.1007/s00701-011-1036-z. Epub 2011 May 8. PMID 21553318
- [Background] Coenen VA, Madler B, Schiffbauer H, Urbach H, Allert N. Individual fiber anatomy of the subthalamic region revealed with diffusion tensor imaging: a concept to identify the deep brain stimulation target for tremor suppression. Neurosurgery. 2011 Apr;68(4):1069-75; discussion 1075-6. doi: 10.1227/NEU.0b013e31820a1a20. PMID 21242831
- [Background] Tomlinson CL, Stowe R, Patel S, Rick C, Gray R, Clarke CE. Systematic review of levodopa dose equivalency reporting in Parkinson's disease. Mov Disord. 2010 Nov 15;25(15):2649-53. doi: 10.1002/mds.23429. PMID 21069833
- [Background] Patel DM, Walker HC, Brooks R, Omar N, Ditty B, Guthrie BL. Adverse events associated with deep brain stimulation for movement disorders: analysis of 510 consecutive cases. Neurosurgery. 2015 Mar;11 Suppl 2(Suppl 2):190-9. doi: 10.1227/NEU.0000000000000659. PMID 25599204
- [Background] Deuschl G, Bain P, Brin M. Consensus statement of the Movement Disorder Society on Tremor. Ad Hoc Scientific Committee. Mov Disord. 1998;13 Suppl 3:2-23. doi: 10.1002/mds.870131303. PMID 9827589
- [Derived] Reinacher PC, Amtage F, Rijntjes M, Piroth T, Prokop T, Jenkner C, Katzler J, Coenen VA. One Pass Thalamic and Subthalamic Stimulation for Patients with Tremor-Dominant Idiopathic Parkinson Syndrome (OPINION): Protocol for a Randomized, Active-Controlled, Double-Blinded Pilot Trial. JMIR Res Protoc. 2018 Jan 30;7(1):e36. doi: 10.2196/resprot.8341. PMID 29382631
- [Derived] Coenen VA, Rijntjes M, Prokop T, Piroth T, Amtage F, Urbach H, Reinacher PC. One-pass deep brain stimulation of dentato-rubro-thalamic tract and subthalamic nucleus for tremor-dominant or equivalent type Parkinson's disease. Acta Neurochir (Wien). 2016 Apr;158(4):773-781. doi: 10.1007/s00701-016-2725-4. Epub 2016 Feb 15. PMID 26876564